CLINICAL TRIAL: NCT06610994
Title: Investigation of the Acute Effect of Local Vibration Application on Gait and Balance in Stroke Patients
Brief Title: Acute Effect of Local Vibration in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, associate professor, Kırıkkale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LocalVibrationStroke
Record Dates: First submitted 2024-05-29; First posted 2024-09-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2024-11

CONDITIONS: Acute Effect of Local Vibration Application in Stroke Patients
Keywords: local vibration; stroke; gait; balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- local vibration apply group (Experimental): Local vibration (LV) application will be made with the Vibrasens© (Techno Concept, Mane, France) device. It will be applied to the most swollen part of the spastic medial gastrocnemius muscles for 10 minutes. LV will be applied to one of the treatment groups at a frequency of 80Hz with an amplitude of 1 mm.
  Interventions: Device: local vibration apply
- placebo group (Placebo Comparator): The device will be contacted to the same areas of the patients in the vibration group for only 10 minutes.
  Interventions: Device: local vibration apply

INTERVENTIONS:
Device: local vibration apply — Local vibration (LV) application will be made with the Vibrasens© (Techno Concept, Mane, France) device. Vibrasens© is a mechanical vibrator that produces transcutaneous vibration stimulations used in sensory-motor rehabilitation. Vibrasens©; It is a non-invasive, therapeutic device. Vibrasens© includes 1 pilot unit, 1 manual vibrator VB200, 4 flat skin contactors for tendon application, 4 round skin contactors for skin application, 1 power supply, 1 user manual and 1 protocol guide. LV application will be applied to the most swollen part of the spastic medial gastrocnemius muscles in the treatment group for 10 minutes. LV will be applied to one of the treatment groups at a frequency of 80Hz with an amplitude of 1 mm.

SUMMARY:
The aim of the research is to examine the acute effect of local vibration application on gait and balance in stroke patients.

DETAILED DESCRIPTION:
The purpose of our study; To examine the acute effect of local vibration application on spatiotemporal parameters of gait and balance in stroke patients.

Many treatment approaches are applied to accelerate motor recovery in stroke rehabilitation. These treatment approaches include Neurodevelopmental Therapy (NGT) treatment approaches and electrotherapy, traditional exercise approaches, as well as new technologies such as robotic devices and virtual reality, which offer new opportunities to increase training intensity by providing a more independent training in the field of rehabilitation. Another treatment approach that has recently attracted attention in neurorehabilitation is local or whole body vibration application. Vibration is defined as "a mechanical stimulus characterized by oscillatory movements". When vibration is viewed biomechanically, it has 3 parameters. These parameters; It is defined as the amplitude that determines the oscillation range of the vibration in millimeters, the frequency that indicates the number of repetitions in one second, and the power given by the acceleration that occurs during vibration.

Vibration can be applied to humans in two basic ways. The first method is local vibration application, which can be applied directly to the muscle or tendon with a hand-held device. The second method, called whole body vibration, is applied on the platform by a vibration source. Vibration applications in physiotherapy are generally 0.1-10 mm amplitude, 10-120 Hz. It is used in frequency and duration from 5 seconds to 60 minutes for up to 72 weeks. In whole body vibration, the degree of acceleration created by the platform surface can create a force up to 17 times the acceleration of gravity.

Wanderley et al. In their study, they applied vibration with a frequency of 100 Hz and an amplitude of 2 mm under the sole of the foot to female patients aged 60 and over with balance problems in 12 sessions of 10-minute applications for 5 weeks. As a result, they reported that vibration stimulation applied to the plantar region had positive effects on postural control and balance in women aged 60 and over with balance problems. In another study, Soffia Naghdi et al. In their case report, they reported that applying 100 Hz frequency plantar vibration to the sole of the foot of a right hemiplegic patient for 5 minutes was effective in balance development. Local vibration, in addition to the general physiotherapy and rehabilitation program, can improve walking performance in patients secondary to chronic stroke. The authors hypothesize that this could possibly be due to mechanical vibration stimulating the brain and reorganizing it. Additionally, the results of another study support this study. It has been shown that after applying low-amplitude local vibration to the flexor carpi radialis muscle and the intrinsic hand muscles of healthy individuals, there is increased excitability in the primary motor cortex area of the stimulated muscle.

When we examined the literature, we could not find any studies investigating the effect of local vibration applications to the gastrocnemius on spatiotemporal parameters and balance of walking in individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years old diagnosed with stroke
* Being diagnosed with ischemic or hemorrhagic stroke,
* Not having cooperation and communication problems,
* Stroke individuals with gastrosoleus spasticity, those with a MAS score of 2 or below,
* Those who score 0-3 on the Modified Rankin Scale.
* People weighing less than 150 kilos
* Patients who can walk independently (with an assisted device if they use an assistive device)

Exclusion Criteria:

* Have undergone surgery or botox for spasticity in the last 6 months,
* Those with joint contracture,
* Having a neurological disease other than stroke that may affect the patient's ability to walk and stand independently, or having pain in the lower extremity joints and a history of fractures in the lower extremities in the last 6 months,
* Having spasticity that prevents sole contact
* Patients who do not agree to participate in the study and do not give written consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 5 minutes
  This scale is a reliable and valid scale that is widely used in the evaluation of muscle tone. Resistance to passive movement is rated from 0 to 4.
Timed Up and Go Test | 5 minutes
  It will be applied for mobility and fall risk. This test will be performed by measuring the time taken by the individual to get up from the chair without arm support after giving the "go" command while sitting in a chair, walking 3 meters in a pre-determined area, turning around and sitting on the chair again without using his or her arms.
Functional Reaching Test | 5 Minutes
  The patient raises his dominant arm 90 degrees, makes a fist, and reaches forward as far as he can to follow the measuring rod placed at shoulder level. Reaching distance is recorded. It is a reliable test with normal values. 15cm and 15cm. Below 15 to 25 cm the risk of falling increases significantly. indicates a moderate fall risk
Biodex Computerized Balance System | 5 minutes
  Individuals' postural control will be evaluated with the Biodex Computerized Balance System. The Biodex Computerized Balance System is a multi-axis device that objectively measures and records an individual's ability to stabilize the relevant joint under dynamic stress. Postural stability test and Fall Risk Test will be performed using two different tests. Postural stability testing evaluates static balance in a standing position. The amount of deviation from the medial-lateral and anterior-posterior axes is calculated as a result of the test. According to these deviation values, general instability index, anterior-posterior stability index and medial-lateral stability index scores are obtained. A fall risk test is a test that objectively evaluates the risk of falling. The reactions of the body according to the changing ground structure are detected and recorded and a value is obtained as a result of the test.
Tandem Stance | 5 minutes
  The test is a test that evaluates static balance in which the area in contact with the ground is narrowed. It is generally preferred in patients who cannot stand on one leg. The patient is asked to stand without support for 30 seconds, with the tip of one foot touching the heel of the other foot. Stopping for less than 10 seconds indicates the risk of falling.
10 Meter Walking Test | 5 minutes
  The 10 meter walk test (10MYT) will be used to measure walking speed. 10MYT is a reliable and valid measurement for measuring walking speed in people who have had a stroke. In this test, the person is asked to walk at his/her normal speed in a pre-measured 10-meter area (if he/she uses a walking aid, it is carried out together with this). The time starts when the person's foot is at the starting line and ends when they cross the finish line. Two measurements are made and the best value is recorded in meters per second (m/s).
Gait Analysis | 10 minutes
  Spatiotemporal parameters of gait will be evaluated using a wireless miniature digital gait analysis system. Gait analysis system is a device that is attached to the person's L5-S1 level with the help of a belt and performs movement analysis in the anteroposterior, mediolateral and superoinferior axes via accelerometer. It transfers the obtained data to the computer via Bluetooth. Sensor: The device is placed in the pelvis at the L5-S1 level over a thin, single layer of clothing. The evaluation will be carried out in a calm environment, with bare feet. Gait parameters evaluated: right and left step lengths, double step length, step width, walking tempo (steps per minute), walking speed and foot angle, pelvic oscillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayvat F, Ozcakar L, Ayvat E, Aksu Yildirim S, Kilinc M. Effects of low vs. high frequency local vibration on mild-moderate muscle spasticity: Ultrasonographical and functional evaluation in patients with multiple sclerosis. Mult Scler Relat Disord. 2021 Jun;51:102930. doi: 10.1016/j.msard.2021.102930. Epub 2021 Mar 31. PMID 33836458
- [Background] Alashram AR, Padua E, Romagnoli C, Annino G. Effectiveness of focal muscle vibration on hemiplegic upper extremity spasticity in individuals with stroke: A systematic review. NeuroRehabilitation. 2019 Dec 18;45(4):471-481. doi: 10.3233/NRE-192863. PMID 31868686
- [Background] Khalifeloo M, Naghdi S, Ansari NN, Akbari M, Jalaie S, Jannat D, Hasson S. A study on the immediate effects of plantar vibration on balance dysfunction in patients with stroke. J Exerc Rehabil. 2018 Apr 26;14(2):259-266. doi: 10.12965/jer.1836044.022. eCollection 2018 Apr. PMID 29740561